CLINICAL TRIAL: NCT06423989
Title: Role of Immunoglobulin in Male Infertility
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Dr Salma kafeel Qureshi (Other)
Responsible Party: Sponsor-Investigator, Dr Salma kafeel Qureshi, Medical director head of Gynaecological and Reproductive unit, Salma Kafeel Medical Centre
Organization: Salma Kafeel Medical Centre (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 102023
Record Dates: First submitted 2024-04-17; First posted 2024-05-21 (Actual); Last update posted 2024-05-21 (Actual); Status verified 2024-05

CONDITIONS: Male Subfertility
MeSH Terms: conditions — Infertility, Male | interventions — Immunoglobulins, Intravenous; pentaglobulin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- male fertility (Experimental)
  Interventions: Combination Product: IVIG

INTERVENTIONS:
Combination Product: IVIG — treatment of subfertility
  Other Names: pentaglobin

SUMMARY:
to investigate the role of IVIG in male infertility and to determine its benefits in term of semen parameters and assisted reproduction outcome

ELIGIBILITY:
Inclusion Criteria:

* male patients

Exclusion Criteria:

* female

Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-04-01 (Actual); Primary Completion 2024-06-01 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
Semen parameters percentage improvement | 6 month
  Sperm concentration/ml
Sperm motility | 6 month
  Percentage active motile sperm
Sperm morphology | 6 month
  Percentage of normal sperm

SECONDARY OUTCOMES:
Assisted Reproduction outcome measure | 12 months
  Percentage of fertilized

CONTACTS AND LOCATIONS:
Locations (1):
- SKMC, Islamabad, Capital, Pakistan

IPD SHARING:
Plan to Share IPD: Yes
with in 6 month
Supporting Information: Study Protocol
Time Frame: 6 month